CLINICAL TRIAL: NCT05758207
Title: Prevalence and Types of Oral Complications Occuring in Hematological Malignancy Patients.:Cross Sectional Study
Brief Title: Oral Complications in Hematological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merit Rafeek Gerges Botros, Assistant lecturer, Assiut University
Other Study IDs: Hematology malignancies
Record Dates: First submitted 2023-02-17; First posted 2023-03-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-05

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The aim of this study was to evaluate the prevalence and types of oral complications found in patients diagnosed with haematological malignancy

DETAILED DESCRIPTION:
Oral lesions can be the first presentation of hematological malignancy. Dentists occasionally are the first healthcare provider that detect oral signs related to a systemic condition and thus contribute to the early diagnosis of the disease 1. Oral health can impact the progression and the outcome of haematological malignancy patients', many patients may suffer from oral infections that might affect hospital stay, treatment cost and patient prognosis 2. The oral manifestations of patients with hematological malignancy can occur due to the disease itself or as a consequence of treatment 3.

Anemia (paleness of mucosa), coagulation disorder, oral petechiae or ecchymosis, spontaneous gingival bleeding and oral infection (Ulcers and overgrowth) may be an oral manifestation of a hematologic malignancy either at diagnosis or during follow up as well as in relapse 4. The treatment of hematologic malignancy includes chemotherapy, radiotherapy, and hematopoietic stem cell transplantation (HSCT). Malignant cells are the target of antineoplastic drugs, but the oral epithelium and other cells with high mitotic rates are usually affected by the treatment. Chemotherapy and the conditioning regimen for HSCT have many adverse effects on the oral tissues depending on the type and dosage of medications 4. Oral mucositis, a common side effect of chemotherapy, causes severe pain, which is only relieved by opioids. Mucositis may appear as a generalized erythema and evolve into painful pseudomembranous ulcers. Neutropenia and thrombocytopenia are also common adverse effects of treatment, leaving patients more susceptible to oral bleeding, infections, and ulcerations. Oral mucosa pigmentation can also occur as an adverse effect of treatment 5. Considering these factors and lack of existing information, a study was designed to investigate the prevalence of oral complications problems occurring in a population of hematological malignancy patients in Assiut University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed patients elder than 18 years with hematological malignancy start from January 1st 2022 to January 1st 2023 including Acute myeloid leukemia Acute lymphoblastic leukemia Chronic myeloid leukemia Chronic lymphoblastic leukemia Non-Hodgkin lymphoma Hodgkin lymphoma Multiple myeloma

Exclusion Criteria:

* Patient younger than 18 years old Patients previously diagnosed Patients refused to participate in our study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed patients elder than 18 years with hematological malignancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Calculate the prevalence of oral complications. | Baseline
  Calculate the prevalence of oral complications with special attention to infectious complications in hematological malignancy patients.

SECONDARY OUTCOMES:
the morbidity related to oral complication in haematological malignancy patients. | Baseline
  Study the morbidity related to oral complication in haematological malignancy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Fayek, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Emodi O, Ohayon C, Bilder A, Capucha T, Wolff A, Rachmiel A. Postextraction Mucormycosis in Immunocompromised-Patient Management and Review of Literature. J Oral Maxillofac Surg. 2021 Jul;79(7):1482-1491. doi: 10.1016/j.joms.2021.01.019. Epub 2021 Jan 25. PMID 33617788
- [Background] Elad S, Zadik Y, Yarom N. Oral Complications of Nonsurgical Cancer Therapies. Atlas Oral Maxillofac Surg Clin North Am. 2017 Sep;25(2):133-147. doi: 10.1016/j.cxom.2017.04.006. No abstract available. PMID 28778303